CLINICAL TRIAL: NCT03366077
Title: A Double-blinded, Randomized, Placebo-controlled, Parallel-group Study Evaluating the Effect of the Probiotic on Recurrent Urinary Tract Infection (UTI) in Adult Women Recently Treated for UTI.
Brief Title: Evaluating the Effect of the Probiotic on Recurrent Urinary Tract Infection in Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CSUB0144
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Urinary Tract Infection in Adult Women
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: double-blinded, randomized, placebo-controlled, parallel-group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): L reuteri
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic

SUMMARY:
Urinary tract infections (UTIs) are the most common bacterial infections in women, with about 50% of women experiencing at least one UTI in their lifetime.

The main pharmacological treatments of cystitis usually involve the use of antibiotics, in particular quinolones (such as ciprofloxacin and levofloxacin), fosfomycin, second-generation and third-generation cephalosporins, and b-lactam antibiotics associated with b-lactamase inhibitors.

DETAILED DESCRIPTION:
This is a double-blinded, randomized, placebo-controlled, parallel-group study evaluating the effect of the probiotic on recurrent urinary tract infection (UTI) in adult women recently treated for UTI.

Primary objective The primary objective is to evaluate the effect of oral supplementation with probiotic on the frequency of UTI during six months from start of intervention in adult women with recurrent UTI.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent for participation in the study.
2. Woman aged 18-50 years old at screening.
3. BMI ≥18 at screening.
4. Currently on antibiotic treatment for UTI, at the time of screening. Antibiotic treatment must stop within three days prior to first IP dose.
5. Recurrent UTI defined as at least two UTIs during the last six months or at least three UTIs during the last 12 months, according to information given by the subject.
6. Able and willing to comply with the restrictions defined for the the study period (see Section 10.6).
7. Access to Bank ID and ability to use the e-health platform (i.e. Internet access).
8. Ability to understand and comply with the requirements of the study, as judged by the Investigator.

Exclusion Criteria:

1. Postmenopausal (defined as 12 months of amenorrhoea).
2. Pregnant or breastfeeding.
3. Planning to become pregnant during the study.
4. Irregular menstruations combined with perimenopausal symptoms.
5. Known hypersensitivity or allergy to any of the components of the test product, or to the comparator (placebo).
6. Use of spermicide contraceptives including spermicidal condom within three days prior to first IP dose.
7. History of complicated cystitis, urgency incontinence, recent pyelonephritis, urological and/or gynaecologist abnormalities, immunocompromised, as judged by the Investigator.
8. Unstable bowel disorder such as diarrhoea, Crohn's disease, ulcerative colitis.

   -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healty women
Enrollment: 140 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rein-Hedin, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One of the participants randomised to the placebo group did not start the intervention, therefore it is a discrepancy between the planned and actual number of started participants.
Groups:
- Active: Probiotics
- Placebo: Placebo control group
Period: Overall Study
Arm/Group | Active | Placebo
Started | 70 | 69
Completed | 61 | 65
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Customized [Mean (Standard Deviation); unit: years] | 30.1 (8.0) | 31.2 (9.3) | 30.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 132
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 64 | 64 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 65 | 67 | 132
Height [Mean (Standard Deviation); unit: cm] | 166.4 (5.4) | 167.2 (6.5) | 166.8 (5.9)
weight [Mean (Standard Deviation); unit: kg] | 65.7 (10.9) | 66.2 (12.7) | 65.9 (11.8)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (3.7) | 23.7 (4.4) | 23.7 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Effect of Oral Supplementation With Lactobacillus Reuteri on the Frequency of Confirmed UTI in Adult Women With Recurrent UTI.
Description: Mean number (Standard Deviation) of confirmed UTIs in adult women with recurrent UTI, during six months from start of intervention, as compared to placebo.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of unique UTIs during study
Groups:
- Active: Sachet 1 - instant drink: Xylitol, Monosodium Citrate, Cranberry Aroma, Cranberry Extract, Grape-skin Extract, Xanthan Gum, Acesulfame Potassium and Zinc Gluconate
  Sachet 2 - probiotic mix: Maltodextrin, L. reuteri DSM 16666 and L. reuteri DSM 17938
- Placebo: Sachet 1 - instant drink: Xylitol, Monosodium Citrate, Cranberry Aroma, Grape-skin Extract, Xanthan Gum and Acesulfame Potassium
  Sachet 2 - maltodextrin: Maltodextrin
Arm/Group | Active | Placebo
Number analyzed (Participants) | 65 | 67
Number of unique UTIs during study | 1.2 (1.4) | 1.3 (1.3)

2. Secondary Outcome: To Evaluate the Effect of Oral Supplementation With Lactobacillus Reuteri on the -Frequency of Confirmed UTI -Time to First Relapse of UTI. -Relapse Rate -Assess the Tolerability
Description: Mean number of confirmed UTIs during the three months intervention period, as compared to placebo.
  Mean number of confirmed UTIs during the three months follow-up period, as compared to placebo.
  Mean time from start of intervention to first relapse of UTI, as compared to placebo.
  Proportion of subjects (%) who experienced at least one confirmed UTI during three months from start of intervention, as compared to placebo.
  Proportion of subjects (%) who experienced at least one confirmed UTI during six months from start of intervention, as compared to placebo.
  Occurrence and frequency of Adverse Events (AEs).
Time Frame: 6 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: In this study, the IP is a food supplement and not an investigational medicinal product.
  However, the procedures for monitoring, collecting and reporting of AEs will be the same as for an investigational medicinal product.
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 3/69
Other Adverse Events (participants affected / at risk) | 36/70 | 36/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=70) | Placebo (N=69)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Concussion with brief loss of consciousness.
Spontaneous miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Abortion spontaneous
Endometritis (Infections and infestations) | 0 (0) | 1 (1) — Endometritis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=70) | Placebo (N=69)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (4)
Nasopharyngitis (Infections and infestations) | 12 (15) | 18 (21)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Dust Allergy (Immune system disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 3 (3)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Worsening post surgical pain (General disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
vulvovaginal candidiasis (Infections and infestations) | 2 (3) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Toe infection (Infections and infestations) | 1 (1) | 0 (0)
head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 2 (2)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Vaginosis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Borrelia (Infections and infestations) | 0 (0) | 1 (1)
blood thyroid stimulating hormone increased (Endocrine disorders) | 0 (0) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
musculosceletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
abortion spontaneous (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometritis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03366077/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT03366077/SAP_001.pdf